CLINICAL TRIAL: NCT00156936
Title: An Open-Label, Multi-Center Study to Evaluate the Long-Term Safety of Medisorb® Naltrexone
Brief Title: ALK21-006EXT: Long-term Safety of Medisorb® Naltrexone (VIVITROL®) in Alcohol- or Opioid-dependent Adults (Extension of Study ALK21-006 [NCT01218997])
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Business decision
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard L. Silverman, MD / VP, Clinical Development, Alkermes, Inc.
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ALK21-006EXT
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Results first posted 2010-11-03 (Estimated); Last update posted 2010-11-17 (Estimated); Status verified 2010-11

CONDITIONS: Alcoholism; Opiate Dependence
MeSH Terms: conditions — Alcoholism; Opioid-Related Disorders | interventions — vivitrol; Naltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medisorb naltrexone 380 mg (VIVITROL) (Experimental)
  Interventions: Drug: Medisorb naltrexone 380 mg
- Oral naltrexone to Medisorb naltrexone 380 mg (VIVITROL) (Experimental)
  Interventions: Drug: Oral naltrexone to Medisorb naltrexone 380 mg

INTERVENTIONS:
Drug: Medisorb naltrexone 380 mg — Administered via intramuscular (IM) injection once every 4 weeks. Subjects in this dosing group also received this treatment throughout the base study.
  Other Names: VIVITROL 380 mg; Naltrexone for extended-release injectable suspension
  Arms: Medisorb naltrexone 380 mg (VIVITROL)
Drug: Oral naltrexone to Medisorb naltrexone 380 mg — Subjects in this dosing group received oral naltrexone 50 mg in the base study, but received only Medisorb naltrexone 380 mg in this extension study, administered via IM injection once every 4 weeks.
  Arms: Oral naltrexone to Medisorb naltrexone 380 mg (VIVITROL)

SUMMARY:
This was a multicenter extension of Alkermes' Study ALK21-006 (NCT01218997) designed to assess the long-term safety of repeat monthly doses of naltrexone long-acting injection. All subjects received open-label Medisorb® naltrexone 380 mg (VIVITROL®).

Planned treatment duration was up to 3 years. Alkermes terminated the study for business purposes in December 2006. The median duration of treatment among all subjects in this extension study was 43 weeks.

DETAILED DESCRIPTION:
From the date of successful completion of Study ALK21-006 (base study [NCT01218997])), all subjects, including those who received oral naltrexone during the base study, were given the option to enroll in this extension study.

Study investigators ensured that subjects were opioid-free and did not demonstrate evidence of withdrawal prior to administration of VIVITROL therapy. If the investigator suspected recent clinically significant opioid use, a naloxone challenge test was performed. The naloxone challenge was not performed in a subject presenting clinical signs or symptoms of opioid withdrawal or in a subject whose urine contained opioids.

ELIGIBILITY:
Primary Inclusion Criteria:

* Adults with a diagnosis of alcohol and/or opioid dependence as defined by the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV) who had satisfactorily completed Alkermes' Study ALK21-006 or other qualifying Medisorb naltrexone study
* Willing and able to return for scheduled clinic visits and study assessments
* Had a stable address
* Agreed to use a contraception for the duration of the study and for 1 month following the last dose if of childbearing potential
* Written informed consent

Primary Exclusion Criteria:

* Pregnancy or lactation
* Terminated early from study drug in a previous Medisorb naltrexone clinical trial
* Any finding that, in the view of the investigator, would compromise the ability to fulfill the protocol visit schedule and/or visit requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2004-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at 17 clinical trial study centers in the United States.
Pre-assignment Details: Investigators ensured subjects were opioid-free (ie, had opioid-free urine screening results) prior to initiation of study therapy. For subjects diagnosed with opioid dependence or in whom clinically significant opioid use was suspected, a naloxone challenge test was performed.
Groups:
- Medisorb Naltrexone 380 mg (VIVITROL): Subjects in this dosing group received VIVITROL (Medisorb naltrexone 380 mg) via intramuscular (IM) injection once every 4 weeks throughout the base study and continued on the same regimen throughout this extension.
- Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL): Subjects in this dosing group switched from oral naltrexone 50 mg daily in the base study to receive VIVITROL (Medisorb naltrexone 380) mg via IM injection once every 4 weeks in this extension study.
Period: Overall Study
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL)
Started | 92 | 16
Completed | 20 | 5
Not Completed | 72 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL) | Total
Number analyzed (Participants) | 92 | 16 | 108
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 92 | 16 | 108
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 42.3 (10.0) | 45.3 (11.5) | 42.7 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 5 | 35
  Male | 62 | 11 | 73
Region of Enrollment [Number; unit: participants]
  United States | 92 | 16 | 108

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Reported at Least 1 Treatment-emergent Adverse Event (TEAE) While on Study.
Description: A TEAE is any adverse event (AE), whether or not considered drug-related, that develops or worsens in severity after study drug administration begins (ie, from the first administration through the end of the follow-up period).
Time Frame: Up to 3 years
Population: Safety population includes all enrolled subjects who received at least 1 dose of study drug (VIVITROL 380 mg) in this extension study.
Measure: Number; unit: Participants
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL)
Number analyzed (Participants) | 62 | 11
Participants | 62 | 11

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years
Description: Safety parameters, including assessment for adverse events (AEs), were conducted at each study visit. All AE reports, whether volunteered, elicited, or observed, were recorded on the appropriate case report forms (CRFs). The recording of AEs began from the time of study enrollment until 30 days after the last dose of study drug.
Arm/Group | Medisorb Naltrexone 380 mg (VIVITROL) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL)
Serious Adverse Events (participants affected / at risk) | 9/92 | 2/16
Other Adverse Events (participants affected / at risk) | 62/92 | 11/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=92) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL) (N=16)
Alcohol dependence syndrome (Psychiatric disorders) | 1 | 0
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Bronchitis acute NOS (Infections and infestations) | 1 | 0
Bronchospasm NOS (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Convulsions NOS (Nervous system disorders) | 1 | 0
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Overdose NOS (Injury, poisoning and procedural complications) | 2 | 0
Pneumonia bacterial NOS (Infections and infestations) | 1 | 0
Pneumonia streptococcal (Infections and infestations) | 1 | 0
Respiratory failure (excl. neonatal) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Staphylococcal infection NOS (Infections and infestations) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Medisorb Naltrexone 380 mg (VIVITROL) (N=92) | Oral Naltrexone to Medisorb Naltrexone 380 mg (VIVITROL) (N=16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Depression (Psychiatric disorders) | 7 | 1
Fatigue (General disorders) | 6 | 1
Headache NOS (Nervous system disorders) | 6 | 1
Nasopharyngitis (Infections and infestations) | 9 | 2
Nausea (Nervous system disorders) | 4 | 2
Toothache (Gastrointestinal disorders) | 6 | 1
Upper respiratory infection (Infections and infestations) | 8 | 2
Influenza (Infections and infestations) | 1 | 2
Sinusitis NOS (Infections and infestations) | 2 | 1
Gastroenteritis viral NOS (Infections and infestations) | 1 | 1
Respiratory tract infection NOS (Infections and infestations) | 1 | 1
UTI (Infections and infestations) | 1 | 1
Urinary tract infection NOS (Infections and infestations) | 1 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Lymph gland infection (Infections and infestations) | 0 | 1
Otitis externa NOS (Infections and infestations) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 1 | 1
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 0 | 1
Leg pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Shoulder bursitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Irritability (Psychiatric disorders) | 1 | 1
Depressive symptom (Psychiatric disorders) | 0 | 1
Transient disorder of initiating or maintaining sleep (Psychiatric disorders) | 0 | 1
Gastritis alcoholic (Gastrointestinal disorders) | 1 | 1
Eructation (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Dizziness (Nervous system disorders) | 3 | 1
Light headedness (Nervous system disorders) | 0 | 1
Mental impairment NOS (Nervous system disorders) | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Weight loss (Investigations) | 2 | 1
Liver function tests NOS abnormal (Investigations) | 1 | 1
Electrocardiogram PR shortened (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Chest pain (General disorders) | 1 | 1
Injection site fibrosis (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Pain NOS (General disorders) | 0 | 1
Post procedural pain (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Limb injury NOS (Injury, poisoning and procedural complications) | 0 | 1
Appetite decreased NOS (Metabolism and nutrition disorders) | 1 | 1
Appetite increased NOS (Metabolism and nutrition disorders) | 0 | 1
Amenorrhea (Reproductive system and breast disorders) | 0 | 1
Menstrual cramps (Reproductive system and breast disorders) | 0 | 1
Sexual dysfunction NOS (Reproductive system and breast disorders) | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 2 | 1
Bruising (Skin and subcutaneous tissue disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Lung nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tympanic membrane hyperaemia (Ear and labyrinth disorders) | 0 | 1
Tympanic membrane perforation (Ear and labyrinth disorders) | 0 | 1
Upper respiratory tract infection NOS (Infections and infestations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should a PI wish to disclose results, the sponsor will review the results communications prior to public release and can embargo results communications for a period of at least 30 days but less than or equal to 90 days from the time submitted to the sponsor for review. Revisions will be negotiated in good faith. For a multicenter study, the institution/PI agree to publish/publicly present the results together with the other sites unless the sponsor grants written permission in advance.